CLINICAL TRIAL: NCT06895902
Title: Suture Eyelid Spring for Eyelid Closure in Patients With Facial Nerve Palsy
Brief Title: Suture Lid Spring for Lid Closure in Patients With Facial Nerve Palsy
Acronym: SESPL
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00149272
Record Dates: First submitted 2025-02-24; First posted 2025-03-26 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Facial Nerve Palsy; Corneal Exposure; Paralytic Lagophthalmos
Keywords: Paralytic lagophthalmos
MeSH Terms: conditions — Bell Palsy; Lagophthalmos

STUDY DESIGN:
Intervention Model Description: non-masked surgical intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Placement of suture lid spring (Experimental): Instead of tying tissue with the surgical suture (polypropylene) that is normally used in lid surgery we will make a loop out of the suture and place it underneath the eyelid skin to see if it will help with eyelid closure in patients with facial nerve palsy.
  There is no placebo or comparison group
  Interventions: Device: Polypropylene Suture Eyelid Spring for Paralytic Lagophthalmos

INTERVENTIONS:
Device: Polypropylene Suture Eyelid Spring for Paralytic Lagophthalmos — The polypropylene loop eyelid suture spring will be centrally placed without fixation to the bone unlike a metal lid spring.

SUMMARY:
The eyelids protect the cornea and eyelid closure is essential to ocular health and clear vision.

Patients with permanent Bells palsy or facial nerve palsy from other reasons such as tumours or trauma may be unable to blink and protect their cornea.

Irreversible visual loss can occur if the cornea is not kept lubricated.

Current treatment options for patients whose eyelid blink does not recover include lubricating the eye every hour or two with drops and lubricating ointment at night, patching the eye closed, sewing parts of the eyelid together (tarsorrpahy), upper lid gold weight or a dental wire spring.

It is inconvenient to lubricate the cornea constantly, and the lubricating drops and ointment usually cost more than $80.00 per month. Lubrication often blurs vision, because the patient must look through a film.

Patching the eye closed and tarsorraphy deprives the patient of peripheral vision, can impede social interaction, and is objectionable cosmetically.

Upper-lid gold weights can be placed underneath the eyelid skin and work by gravity. A gold weight will only work when the patient initiates a forced blink. Gold weights may not work when the patient is lying down because there is no gravity to assist lid closure. The eyelid skin is the thinnest skin in the body and can extrude through the skin over time.

Eyelid springs made of metal dental wire exist but are not frequently used because they often extrude through the thin eyelid skin. Also, dental wire springs require attachment to the bone near the side of the eye. It is not uncommon that dental wire springs have to be removed or replaced.

The investigators propose a new spring to close the eyelid made out of the surgical stitches (sutures) commonly used in medicine and eyelid surgery. The stitch will be made into a custom shape and attached underneath the skin near the centre of the lid, without attachment to the bone.

Upper lid gold weights, dental wire springs, and our proposed suture spring are all foreign bodies and can all become infected or extrude through the skin. Because the suture spring is thinner than a gold weight and because it does not have sharp edges like a metal spring, there should be less risk of extrusion. The suture spring will lose its elasticity over time and will require replacement.

DETAILED DESCRIPTION:
PURPOSE: To develop and test a plastic lid spring to help patients with facial nerve palsy who cannot close their eyes (paralytic lagophthalmos) and protect their cornea.

HYPOTHESIS: Polypropylene monofilament suture (Prolene) is Health Canada-approved and commonly used in surgery including surgery in the eyelid region. When the prolene suture is coiled in a loop it has elastic spring that can assist in lid closure. If the prolene loop coil is sutured to the tarsus and underneath the orbital septum inferior to the superior orbital rim, it should help keep the eyelid closed, while still allowing the levator and Mullers muscles to open the lid.

JUSTIFICATION: Current methods to help patients with paralytic lagophthalmos require improvement. Tarsorraphy decreases peripheral vision and adversely affects cosmesis. Gold weights are static and require a forced blink and gravity to work. Gold weights may not help when the patient is supine. Wire lid springs require suturing or fixation to the lateral orbital bone and extensive dissection. The thin dental wire frequently extrudes through the skin.

In contrast to the above a plastic suture lid spring would be placed in the central lid with less dissection than a dental wire spring, and about the same amount of dissection as a gold weight. As the plastic has innate elasticity it provides dynamic lid closure whether the patient is upright or supine.

OBJECTIVES AND METHOD:

1. FORCE DETERMINATION

   The amount of force required to close the lids is estimated by F=m*g, where m is in the range of 1.2 to 1.4 grams and g is 9.81 m/s^2. The investigators will measure the dynamic force of 10 mm compression on the prolene suture. Ten mm is the sum of normal vertical palpebral fissure height (margin reflex distance 1 and margin reflex distance 2.) Prolene suture loops of calibres from 5-0 to 2 will be tested in a mechanical engineering laboratory. Since humans may blink 12 times per minute of the waking day, repetitive strain tests will be performed to determine the longevity of the plastic spring.
2. CADAVER STUDY

   The cadavers will be accessed through the University of Alberta anatomy lab, general surgery anatomy service and used in keeping with the intent of the donors and donor families. The investigators will not be collecting identifiers.

   A 2 mm deep incision will be made in the upper eyelid, 2 centimeters in length. The investigators will place the prolene suture in the cadaver lid underneath the septum superiorly and suture to the tarsus inferiorly. The cadaver study will allow optimal determination of the anatomic placement of the suture for human studies. The prolene loop can be custom-sized for the wound bed and tied to itself once the desired size is achieved.
3. HUMAN STUDIES

Patients with lagophthalmos will have short to long-term placement of the prolene loop. Because of the local anesthetic, and bleeding and bruising, approximately 1 month will be required to determine if the prolene loop is beneficial, or whether it should be removed and a gold weight implanted instead. During this 1 month the patient with paralytic lagophthalmos is not at any increased risk of corneal exposure than during their pre-operative state and should maintain their corneal lubrication.

As there are only a limited number of patients with paralytic lagophthalmos, further testing can be performed on ptosis patients undergoing anterior levator Patients with anterior ptosis repair will have temporary placement of the lid spring, and blink dynamics will be observed. Note that patients requiring ptosis repair have the same anatomic dissection as required for the plastic spring. The placement of the prolene spring will in no way harm the result of the ptosis surgery. The prolene plastic spring will be placed for about 2 minutes to observe blink dynamics and removed and the ptosis surgery will proceed as usual.

In the patients with paralytic lagophthalmos. Pre-operative lagophthalmos in mm, House-Brackman score for facial nerve impairment, visual acuity, corneal status, corneal sensation, Bells phenomenon, lid contour and cosmesis, will be recorded. The same measurements will be repeated at the post-operative 1 week, 1-month, 2-month, 6-month, and 12-month checks.

PLAN FOR DATA ANALYSIS

Paired t-tests will be used to compare the pre-operative and 1-month post-operative results, and then to compare the 1 month with the 6-month results.

The investigators will monitor the patients over a 12-month period to see if the lid spring loses elasticity or has wound complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older with facial nerve transection or paralytic lagophthalmos that has not improved after 6 weeks.

Exclusion Criteria:

* Patients unable to tolerate awake eyelid surgery under local anesthetic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | within the first 2 weeks.
  Amount of lid closure in millimetres

CONTACTS AND LOCATIONS:
Overall Officials: Edsel Ing, MD PhD FRCSC, Principal Investigator — University of Alberta
Locations (1):
- Eye Institute of Alberta, Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No